CLINICAL TRIAL: NCT01391182
Title: Epsilon Aminocaproic Acid (EACA) for the Reduction of Blood Loss in Total Hip Arthroplasty (THA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mary O'Connor, Chair, Department of Orthopedic Surgery, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 11-001111
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Degenerative Joint Disease; Osteoarthritis
Keywords: Epsilon Aminocaproic Acid; blood loss; total hip arthroplasty; reduction in blood transfusions; Amicar
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EACA arm (Active Comparator): In order to obtain sufficient power, a total of 120 patients will be studied, 60 in each group. The surgeon performing the case, their staff, the anesthesiologist, nurse anesthetist and the patient will be blinded to whether the patient received EACA or placebo. Pharmacy will prepare the EACA dose or the saline. Serum hemoglobin levels with be drawn preoperatively and on post operative days one, two, and three. The first dose will be given in the operating room prior to incision (within 30 minutes of the incision). The second dose will be given four hours after the first dose. Two doses are given due to the short half-life of EACA. The timing of administration of EACA will be recorded.
  Interventions: Other: EACA
- Placebo arm (Placebo Comparator): In order to obtain sufficient power, a total of 120 patients will be studied, 60 in each group. The surgeon performing the case, their staff, the anesthesiologist, nurse anesthetist and the patient will be blinded to whether the patient received EACA or placebo. Pharmacy will prepare the EACA dose or the saline. Serum hemoglobin levels with be drawn preoperatively and on post operative days one, two, and three. The first dose will be given in the operating room prior to incision (within 30 minutes of the incision). The second dose will be given four hours after the first dose. Two doses are given due to the short half-life of EACA. The timing of administration of EACA will be recorded.
  Interventions: Other: Placebo arm

INTERVENTIONS:
Other: EACA — EACA 5 grams IV (mixed in NS) given in two doses: prior to incision (total hip arthroplasty) and repeated 4 hours later.
  Arms: EACA arm
Other: Placebo arm — Placebo (NS) IV given in two doses: prior to incision (total hip arthroplasty) and repeated 4 hours later.
  Arms: Placebo arm

SUMMARY:
You are being asked to take part in this research study because you are scheduled to have total hip replacement (arthroplasty) surgery. The goal of this study is to evaluate the effectiveness of the drug, epsilon Aminocaproic Acid (EACA), in decreasing the need for patients to receive blood after surgery. Currently, EACA is approved by the Federal Drug Administration (FDA) to treat a patient who is bleeding. The investigators plan to use EACA to prevent bleeding during and after surgery; use of this drug as a means of preventing bleeding is not currently approved by the FDA.

DETAILED DESCRIPTION:
The goal of this prospective randomized study is to evaluate the effectiveness of a drug, epsilon aminocaproic acid (EACA), in reducing the frequency of postoperative blood transfusion following primary total hip arthroplasty. In our institution, up to 40% of patients with a preoperative of 13.5 g/dl or less undergoing total hip arthroplasty will require a blood transfusion. Fibrinolytic drugs such as EACA and tranexamic acid (TA) have been shown to decrease blood loss during surgery and decrease the likelihood of blood transfusion during postoperative hospitalization.. Both drugs decrease the body's ability to break down a blood clot, thus pushing the balance of blood clot formation and breakdown towards clot formation. This mechanism can decrease the amount of blood loss during and after a surgical procedure. The haemostatic effect of EACA has been investigated in multiple studies with the majority showing a positive effect on postoperative hemoglobin levels and decreased blood transfusion rates. Though several studies exist revealing the effective and safe use of perioperative TA, a similar drug to EACA, there is a paucity of information on the use of EACA in total joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for a primary total hip arthroplasty to be performed at the Mayo Clinic
2. A preoperative hemoglobin between 10.0 and 13.5

Exclusion Criteria:

1. A preoperative hemoglobin less than 10.0 or greater than 13.5
2. Revision arthroplasty;
3. Arthroplasty performed for acute fracture
4. Inability to obtain informed consent;
5. Allergy to EACA
6. Pregnancy
7. History of coronary stenting < 6 months
8. Heart valve replacement;
9. Renal disease,
10. Coagulopathy, DIC,
11. embolic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin levels and transfusion rates. | 96 hours after total hip arthroplasty surgery.
  Postoperative hemogloblins will be monitored on postop day 1, 2, and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Mary I O'Connor, MD, Principal Investigator — Mayo Clinic Jacksonville, Chair, Orthopedics
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States